CLINICAL TRIAL: NCT05932966
Title: Comparison With Observational Methods and Performance Assessment From Real-life Experience of Closed-Loop Insulin Delivery Systems
Acronym: COMPARE-CLIDS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/0024
Record Dates: First submitted 2023-06-21; First posted 2023-07-06 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes type 1; closed loop insulin delivery system; continuous glucose monitoring; sensor-augmented pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with type 1 Diabetes equipped with control-IQ closed loop system: Patients with type 1 Diabetes equipped with control-IQ closed loop system
  Interventions: Device: Insulin closed-loop delivery system
- Patients with type 1 diabetes equipped with Smart GUARD closed loop system: Patients with type 1 diabetes equipped with Smart GUARD closed loop system
  Interventions: Device: Insulin closed-loop delivery system

INTERVENTIONS:
Device: Insulin closed-loop delivery system — Insulin closed-loop delivery system

SUMMARY:
This study aims to compare glycemic control obtained under closed loop depending on the system : Smartguard (Medtronic 780) versus Control IQ (Tandem) in patients with diabetes type 1.

DETAILED DESCRIPTION:
Since 2021, several closed-loop insulin delivery systems have been reimbursed in France for patients living with type 1 diabetes. The "real-life" efficacy and safety of these systems have already been the subject of several publications, confirming the results of clinical trials.

To date, there are no clinical trial comparing closed-loop systems. There are, however, a few observational studies that have attempted such a comparison, but with few patients included or a poorly adapted methodology.

Given the size of the cohort of patients with type 1 diabetes fitted with a closed-loop system in the diabetology department of the Centre Hospitalier Sud-Francilien since 2021 (> 400), we propose a single-center analysis to compare real-life performance of Smartguard (Medtronic 780) versus Control IQ (Tandem) in patients with diabetes type 1 during a follow-up of 12 months and using a propensity score

ELIGIBILITY:
Inclusion Criteria:

* Patient > 16 years
* Patient with diabetes type 1.
* Patient treated with a CONTROL-IQ or SMARTGUARD closed-loop insulin delivery system between 01/2021 and 05/2022.
* Follow-up patient in Centre Hospitalier Sud Francilien

Exclusion Criteria:

* Women who had pregnancy within 12 months of system initiation.
* Patient who have been treated with both systems within 12 months.
* Patient or parental authority objecting the use of data

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The population will be selected from the diabetes department of a French public hospital. All eligible patients will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Comparison of glycemic control obtained under closed loop according to the system used: SG versus CIQ | at 12 months
  Time spent in target range (between 70 and 180 mg/dL) after 12 months following initiation of the closed-loop system, as measured by continuous glucose monitoring (CGM).system, as measured by continuous glucose monitoring (CGM).

SECONDARY OUTCOMES:
Time below target (< 70 mg/dL) | at 12 months
  Compare glycemic control
Glycemic coefficient of variation (CV) | at 12 months
  Compare glycemic control
glucose management indicator | at 12 months
  Compare glycemic control
HBA1c | at 12 months
  Compare glycemic control
weight daily insulin dose | at 12 months
  Compare glycemic control
daily insulin dose | at 12 months
  Compare glycemic control

CONTACTS AND LOCATIONS:
Overall Officials: Coralie AMADOU, PHD, Principal Investigator — Centre Hospitalier Sud Francilien
Locations (1):
- Centre Hospitalier Sud Francilien, Corbeil-Essonnes, France

IPD SHARING:
Plan to Share IPD: No